CLINICAL TRIAL: NCT05688085
Title: A Randomized, Open-label, Crossover, Phase 1 Study to Evaluate Pharmacokinetics and Safety of Irbesartan High/Amlodipine Fixed Dose Combination in Comparison With Co-administration of Mono Compounds in Healthy Volunteers
Brief Title: Pharmacokinetics of Irbesartan High/Amlodipine FDC and Co-administration of Irbesartan High and Amlodipine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HD-AI-103
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irbesartan High/Amlodipine Fixed dose combination (Experimental): participants will receive one tablet of Irbesartan High/Amlodipine FDC in a crossover design
  Interventions: Drug: Irbesartan High/Amlodipine FDC
- Co-administration of Irbesartan High and Amlodipine (Experimental): participants will receive one table each of Irbesartan High and Amlodipine in a crossover design
  Interventions: Drug: Irbesartan High; Drug: Amlodipine

INTERVENTIONS:
Drug: Irbesartan High/Amlodipine FDC — Irbesartan High/Amlodipine FDC
  Arms: Irbesartan High/Amlodipine Fixed dose combination
Drug: Irbesartan High — Co-administration of Irbesartan High and Amlodipine
  Arms: Co-administration of Irbesartan High and Amlodipine
Drug: Amlodipine — Co-administration of Irbesartan High and Amlodipine
  Arms: Co-administration of Irbesartan High and Amlodipine

SUMMARY:
The purpose of this study is to compare pharmacokinetics and safety of Irbesartan High and Amlodipine Fixed Dose Combination and coadministration of mono compounds in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older on screening
* Signed informed consent
* Healthy Volunteer
* Other inclusion applied

Exclusion Criteria:

* Clinically relevant/significant findings as evaluated by the investigator
* Other exclusion applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
AUCt of Irbesartan High and Amlodipine | 72 hours
Cmax of Irbesartan High and Amlodipine | 72 hours

SECONDARY OUTCOMES:
AUCinf of Irbesartan High and Amlodipine | 72 hours
AUCt/AUCinf of Irbesartan High and Amlodipine | 72 hours
tmax of Irbesartan High and Amlodipine | 72 hours
half-life of Irbesartan High and Amlodipine | 72 hours
CL/F of Irbesartan High and Amlodipine | 72 hours
Vz/F of Irbesartan High and Amlodipine | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea